CLINICAL TRIAL: NCT01835145
Title: Randomized Phase II Study Comparing the MET Inhibitor Cabozantinib to Temozolomide/Dacarbazine in Ocular Melanoma
Brief Title: Cabozantinib-S-Malate Compared With Temozolomide or Dacarbazine in Treating Patients With Metastatic Melanoma of the Eye That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Exelisis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00821; NCI-2013-00821 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CALGB-A091201; A091201; A091201 (Other: Alliance for Clinical Trials in Oncology); A091201 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Recurrent Uveal Melanoma; Stage III Uveal Melanoma AJCC v7; Stage IIIA Uveal Melanoma AJCC v7; Stage IIIB Uveal Melanoma AJCC v7; Stage IIIC Uveal Melanoma AJCC v7; Stage IV Uveal Melanoma AJCC v7
MeSH Terms: conditions — Uveal Melanoma | interventions — cabozantinib; Dacarbazine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (cabozantinib-s-malate) (Experimental): Patients receive cabozantinib-s-malate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis
- Arm II (temozolomide or dacarbazine) (Experimental): Patients receive temozolomide PO daily on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. If temozolomide is not available, patients receive dacarbazine IV over 15-60 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dacarbazine; Other: Laboratory Biomarker Analysis; Drug: Temozolomide

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL-184; XL184
  Arms: Arm I (cabozantinib-s-malate)
Drug: Dacarbazine — Given IV
  Other Names: 4-(Dimethyltriazeno)imidazole-5-carboxamide; 5-(Dimethyltriazeno)imidazole-4-carboxamide; Asercit; Biocarbazine; Dacarbazina; Dacarbazina Almirall; Dacarbazine - DTIC; Dacatic; Dakarbazin; Deticene; Detimedac; DIC; Dimethyl (triazeno) imidazolecarboxamide; Dimethyl Triazeno Imidazol Carboxamide; Dimethyl Triazeno Imidazole Carboxamide; dimethyl-triazeno-imidazole carboxamide; Dimethyl-triazeno-imidazole-carboximide; DTIC; DTIC-Dome; Fauldetic; Imidazole Carboxamide; Imidazole Carboxamide Dimethyltriazeno; WR-139007
  Arms: Arm II (temozolomide or dacarbazine)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ
  Arms: Arm II (temozolomide or dacarbazine)

SUMMARY:
This randomized phase II trial studies how well cabozantinib-s-malate works compared with temozolomide or dacarbazine in treating patients with melanoma of the eye (ocular melanoma) that has spread to other parts of the body and cannot be removed by surgery. Cabozantinib-s-malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide and dacarbazine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether cabozantinib-s-malate works better than temozolomide or dacarbazine in treating patients with melanoma of the eye.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the progression-free survival rate at 4 months (PFS4) of patients with ocular melanoma treated with cabozantinib-s-malate (cabozantinib) or temozolomide (or dacarbazine).

SECONDARY OBJECTIVES:

I. Estimate the distribution of progression-free survival (PFS) times. II. Estimate the distribution of overall survival (OS) times. III. Estimate the confirmed response rate as determined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

IV. Assess the safety of these agents by examining the toxicity profile. V. Correlate the response of MET molecular status.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cabozantinib-s-malate orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive temozolomide PO daily on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. If temozolomide is not available, patients receive dacarbazine intravenously (IV) over 15-60 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed uveal melanoma that is metastatic or unresectable; if histologic or cytologic confirmation of the primary is not available, confirmation of the primary diagnosis of uveal melanoma by the treating investigator can be clinically obtained, as per standard practice for uveal melanoma; pathologic confirmation of diagnosis will be performed at the participating site
* Measurable disease defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan or magnetic resonance imaging (MRI)
* Prior systemic therapies allowed, except for those treatments directed toward, or with activity against, c-Met or vascular endothelial growth factor/receptor (VEGF/R), and the chemotherapy agents temozolomide and dacarbazine; prior treatment must have been no earlier than 3 weeks prior to starting treatment with cabozantinib with exceptions noted below and the following: at least 4 weeks since prior hepatic infusion or at least 2 weeks since radiation therapy
* No cytotoxic chemotherapy including investigational cytotoxic chemotherapy or biologic agents (e.g., cytokines or antibodies) within the last 3 weeks, or nitrosoureas/mitomycin C within 6 weeks before the first dose of study treatment; at least 6 weeks must have elapsed if the last regimen included an anti-cytotoxic T-lymphocyte antigen 4 (CTLA4) antibody; patients must have experienced disease progression on their prior therapy in the opinion of the treating investigator
* No prior radiation therapy within the last 4 weeks, except as below

  * To the thoracic cavity, abdomen, or pelvis within 12 weeks before the first dose of study treatment, or has ongoing complications, or is without complete recovery to < grade 1 toxicity
  * To bone or brain metastasis within 14 days before the first dose of study treatment
  * To any other site(s) within 28 days before the first dose of study treatment
  * Prior radiation treatment may have included no more than 3000 centigray (cGy) to fields including substantial bone marrow
* No prior radionuclide treatment within 6 weeks of the first dose of study treatment
* No prior treatment with a small molecule kinase inhibitor or a hormonal therapy within 14 days or 5 half-lives (whichever is longer)
* No concomitant anti-cancer therapy unless specified above
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* A corrected QT interval calculated by the Fridericia formula (QTcF) =< 500 ms within 28 days before randomization; Note: if initial QTcF is found to be > 500 ms, two additional electrocardiograms (EKGs) separated by at least 3 minutes should be performed; if the average of these three consecutive results for QTcF is =< 500 ms, the patient meets eligibility in this regard
* Common Terminology Criteria for Adverse Events (CTCAE) recovered to baseline or CTCAE =< grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant adverse events (AEs)
* No active brain metastases or epidural disease; patients with brain metastases previously treated with whole brain radiation or radiosurgery or patients with epidural disease previously treated with radiation or surgery who are asymptomatic and do not require steroid treatment for at least 2 weeks before starting study treatment are eligible; neurosurgical resection of brain metastases or brain biopsy is permitted if completed at least 12 weeks before starting study treatment; baseline brain imaging with contrast-enhanced CT or MRI scans for patients with known brain metastases is required to confirm eligibility
* No clinically significant gastrointestinal bleeding within 24 weeks before the first dose of study treatment
* No hemoptysis of >= 0.5 teaspoon (2.5 mL) of red blood within 12 weeks before the first dose of study treatment
* No signs indicative of pulmonary hemorrhage within 12 weeks before the first dose of study treatment
* No prior radiographic evidence of cavitating pulmonary lesion(s)
* No tumor in contact with, invading or encasing any major blood vessels
* No evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of treatment
* The patient may not have uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including:

    * Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening
    * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mmHg systolic, or > 90 mmHg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment
    * Any history of congenital long QT syndrome
    * Any of the following within 24 weeks before the first dose of study treatment:

      * Unstable angina pectoris
      * Clinically-significant cardiac arrhythmias
      * Stroke (including transient ischemic attack [TIA], or other ischemic event)
      * Myocardial infarction
      * Thromboembolic event requiring therapeutic anticoagulation (Note: patients with a venous filter [e.g. vena cava filter] are not eligible for this study)
  * Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

    * Any of the following within 28 days before the first dose of study treatment

      * Intra-abdominal tumor/metastases invading GI mucosa
      * Active peptic ulcer disease
      * Inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
      * Malabsorption syndrome
    * Any of the following within 24 weeks before the first dose of study treatment:

      * Abdominal fistula
      * Gastrointestinal perforation
      * Intra-abdominal abscess; Note: complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more that 24 weeks before the first dose of study treatment
      * Bowel obstruction or gastric outlet obstruction
  * Other clinically significant disorders such as:

    * Serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
    * History of organ transplant
    * Concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment
    * History of major surgery as follows:

      * Major surgery in past 8 weeks of the first dose of cabozantinib if there were no wound healing complications or within 24 weeks of the first dose of cabozantinib if there were wound complications
      * Minor surgery within 4 weeks of the first dose of cabozantinib if there were no wound healing complications or within 12 weeks of the first dose of cabozantinib if there were wound complications
      * In addition, complete wound healing from prior surgery must be confirmed at least 28 days before the first dose of cabozantinib irrespective of the time from surgery
    * Active infection requiring systemic treatment within 28 days before the first dose of study treatment
* No concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or factor Xa inhibitors, or antiplatelet agents (e.g., clopidogrel); low dose aspirin (=< 81 mg/day), low-dose warfarin (=< 1 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted; please note that drugs that strongly induce or inhibit cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) or are associated with a risk of Torsades are not allowed; chronic concomitant treatment of CYP3A4 inducers is not allowed (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's wort); as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product; the following drugs are strong inhibitors of CYP3A4 and are not allowed during the treatment with cabozantinib:

  * Boceprevir
  * Indinavir
  * Nelfinavir
  * Lopinavir/ritonavir
  * Saquinavir
  * Telaprevir
  * Ritonavir
  * Clarithromycin
  * Conivaptan
  * Itraconazole
  * Ketoconazole
  * Mibefradil
  * Nefazodone
  * Posaconazole
  * Voriconazole
  * Telithromycin
  * Drugs with possible or conditional risk of torsades should be used with caution knowing that cabozantinib could prolong the QT interval
* Patients who are pregnant or nursing are not eligible; women of child bearing potential must have a negative serum or urine pregnancy test within 16 days prior to registration; women of child-bearing potential include:

  * Any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea >= 12 consecutive months)
  * Women on hormone replacement therapy (HRT) with documented serum follicle stimulating hormone (FSH) level > 35m IU/mL
  * Women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy)
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to cabozantinib, temozolomide and dacarbazine
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 × upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5.0 × institutional upper limit of normal (for patients with metastases); AST (SGOT)/ALT (SGPT) =< 2.5 × institutional upper limit of normal (for patients without metastases)
* Serum creatinine =< 1.5 × ULN, OR calculated creatinine clearance >= 30 mL/minute (modified Cockcroft and Gault formula)
* Hemoglobin >= 9 g/dL
* Serum albumin >= 2.8 g/dL
* Urine protein/creatinine ratio (UPCR) =< 1; if urine/protein creatinine (UPC) >= 1, then a 24-hour urine protein must be assessed; eligible patients must have a 24-hour urine protein value < 1 g/L
* Thyroid-stimulating hormone (TSH) within normal limits (WNL); supplementation is acceptable to achieve a TSH WNL; in patients with abnormal TSH however free T4 and free thyroxine index (FTI) are normal and patient is clinically euthyroid, patient is eligible
* Prothrombin time (PT)/international normalized ratio (INR) must be =< 1.2 x the laboratory ULN
* No clinical or radiographic evidence of pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-07-31 (Actual); Primary Completion 2016-10-21 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Luke, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (228):
- United States (224):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Cox Cancer Center Branson, Branson, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Bao R, Surriga O, Olson DJ, Allred JB, Strand CA, Zha Y, Carll T, Labadie BW, Bastos BR, Butler M, Hogg D, Musi E, Ambrosini G, Munster P, Schwartz GK, Luke JJ. Transcriptional analysis of metastatic uveal melanoma survival nominates NRP1 as a therapeutic target. Melanoma Res. 2021 Feb 1;31(1):27-37. doi: 10.1097/CMR.0000000000000701. PMID 33170593

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Cabozantinib-s-malate): Patients receive 60 mg cabozantinib-s-malate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm II (Temozolomide or Dacarbazine): Patients receive 150 mg/m^2 temozolomide PO daily on days 1-5 of a 28 day cycle. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  If temozolomide is not available, patients receive 1000 mg/m^2/day dacarbazine IV over 15-60 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I (Cabozantinib-s-malate) | Arm II (Temozolomide or Dacarbazine)
Started | 32 | 15
Completed | 31 | 15
Not Completed | 1 | 0
Not completed — Ineligible prior to treatment | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants that began study treatment are included in the baseline analysis.
Groups:
- Arm II (Temozolomide or Dacarbazine): Patients receive 150 mg/m^2 temozolomide PO daily on days 1-5 of a 28 day cycle. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. >>
  >> If temozolomide is not available, patients receive 1000 mg/m^2/day dacarbazine IV over 15-60 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Arm I (Cabozantinib-s-malate) | Arm II (Temozolomide or Dacarbazine) | Total
Number analyzed (Participants) | 31 | 15 | 46
Age, Continuous [Median (Full Range); unit: years] | 60 [30 to 86] | 67 [45 to 78] | 62.5 [30 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 17 | 9 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 31 | 15 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 8 | 3 | 11
  United States | 23 | 12 | 35

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Without a Progression Free Survival Event at 4 Months (PFS4)
Description: A patient will be declared a PFS4 success if they are on study and progression free for at least 4 months. Progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, with an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression. The success for each arm will be calculated independently as the number of successes divided by the total number of evaluable patients. A one-sided chi-squared test for a difference in PFS4 proportions will be used to test for a difference between arms.
Time Frame: At 4 months
Population: All patients that began protocol treatment were included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Arm II (Temozolomide or Dacarbazine): Patients receive 150 mg/m^2 temozolomide PO daily on days 1-5 of a 28 day cycle. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  >
  > If temozolomide is not available, patients receive 1000 mg/m^2/day dacarbazine IV over 15-60 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I (Cabozantinib-s-malate) | Arm II (Temozolomide or Dacarbazine)
Number analyzed (Participants) | 31 | 15
proportion of participants | .323 [.167 to .514] | .267 [.078 to .551]
Statistical Analysis 1: Comparison: Arm I (Cabozantinib-s-malate) vs Arm II (Temozolomide or Dacarbazine); A one-sided chi-squared test for a difference in PFS4 rates will be used to test for a difference between arms; Test type: Superiority; p = 0.70, Chi-squared

2. Secondary Outcome: Confirmed Response Rate as Determined by the RECIST Criteria (Version 1.1)
Description: The confirmed response rates will be estimated by dividing the number of confirmed responders by the number of evaluable patients. 95% confidence intervals will be calculated.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cabozantinib-s-malate) | Arm II (Temozolomide or Dacarbazine)
Number analyzed (Participants) | 31 | 15
Participants | 0 | 0

3. Secondary Outcome: Percentage of Patients Who Experienced Grade 3+ Adverse Events Regardless of Attribution
Description: percentage of patients who experienced grade 3+ adverse events regardless of attribution, graded according to the National Cancer Institute CTCAE version 4.0
Time Frame: Up to 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Arm I (Cabozantinib-s-malate) | Arm II (Temozolomide or Dacarbazine)
Number analyzed (Participants) | 31 | 15
percentage of patients | 51.6 | 20

4. Secondary Outcome: Overall Survival (OS)
Description: The distribution of OS time will be estimated using the method of Kaplan Meier.
Time Frame: Number of days from registration until death, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Cabozantinib-s-malate) | Arm II (Temozolomide or Dacarbazine)
Number analyzed (Participants) | 31 | 15
months | 6.3 [5.5 to 10.3] | 7.2 [5.6 to NA] — The 95% confidence interval upper limit was not estimated (insufficient number of participants with events).

5. Secondary Outcome: PFS
Description: The distribution of PFS time will be estimated using the method of Kaplan Meier and is defined as the number of days from registration until disease progression (or death). Progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, with an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Number of days from registration until disease progression (or death), assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Cabozantinib-s-malate) | Arm II (Temozolomide or Dacarbazine)
Number analyzed (Participants) | 31 | 15
months | 2.0 [1.8 to 5.3] | 1.9 [1.8 to 5.0]

6. Other Pre Specified Outcome: Pre-treatment GNAQ/GNA11 and Potentially Other Mutations in Tissue
Description: The proportions of patients within these groups pre-treatment will be presented with 90% exact binomial confidence intervals. These findings will be correlated with overall survival using a Student's T-test.
Time Frame: Baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Pre-treatment Immune Gene Expression in Tissue Defined as T Cell-inflamed, Intermediate and Non-T Cell-inflamed
Description: as for outcome 6
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Arm II (Temozolomide): Patients receive 150 mg/m^2 temozolomide PO daily on days 1-5 of a 28 day cycle. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm II (Dacarbazine): Patients receive 1000 mg/m^2/day dacarbazine IV over 15-60 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I (Cabozantinib-s-malate) | Arm II (Temozolomide) | Arm II (Dacarbazine)
All-Cause Mortality (participants affected / at risk) | 2/31 | 1/11 | 0/4
Serious Adverse Events (participants affected / at risk) | 15/31 | 6/11 | 2/4
Other Adverse Events (participants affected / at risk) | 30/31 | 11/11 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Cabozantinib-s-malate) (N=31) | Arm II (Temozolomide) (N=11) | Arm II (Dacarbazine) (N=4)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (5) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 4 (4) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Cabozantinib-s-malate) (N=31) | Arm II (Temozolomide) (N=11) | Arm II (Dacarbazine) (N=4)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 6 (9) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (17) | 2 (6) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (5) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (6) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (6) | 3 (6) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 15 (41) | 4 (6) | 2 (5)
Dry mouth (Gastrointestinal disorders) | 4 (5) | 1 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (4) | 2 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (20) | 6 (16) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (2) | 1 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 4 (6) | 1 (3)
Chills (General disorders) | 0 (0) | 1 (3) | 1 (6)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 20 (51) | 10 (31) | 3 (5)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (5) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 21 (71) | 6 (17) | 1 (3)
Alkaline phosphatase increased (Investigations) | 5 (9) | 3 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 26 (85) | 10 (26) | 2 (4)
Blood bilirubin increased (Investigations) | 6 (10) | 3 (4) | 2 (3)
Creatinine increased (Investigations) | 2 (4) | 1 (4) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1)
Hemoglobin increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (3) | 2 (10) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (3) | 3 (7) | 0 (0)
Neutrophil count decreased (Investigations) | 7 (13) | 2 (6) | 2 (5)
Platelet count decreased (Investigations) | 12 (27) | 5 (9) | 2 (6)
Weight loss (Investigations) | 6 (9) | 2 (9) | 0 (0)
White blood cell decreased (Investigations) | 3 (5) | 4 (8) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 7 (14) | 3 (10) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 4 (9) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 3 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (4) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (10) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (6) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (11) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 1 (3) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (3) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 6 (10) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (8) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (5) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (5) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (9) | 1 (1) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (5) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (3) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (3) | 0 (0)
Hypertension (Vascular disorders) | 18 (61) | 5 (17) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (4) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less